CLINICAL TRIAL: NCT03880305
Title: White Blood Cells and Platelets Indices as a Prognostic Factor in Neonatal Sepsis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eslam Ahmad Roshdy, Principal investigator, Assiut University
Other Study IDs: WBCPLATNS
Record Dates: First submitted 2019-03-13; First posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Neonatal Sepsis
Keywords: neonatal sepsis; white blood cells; platelets
MeSH Terms: conditions — Neonatal Sepsis | interventions — Blood Cell Count; Blood Culture

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: complete blood count — complete blood count
  Other Names: blood culture

SUMMARY:
Sepsis is a complex condition initiated by a pathogen and mediated by cytokines followed by immune, inflammatory, and coagulation homeostasis disturbances, its evolution being dictated by a complicated balance between pro inflammatory and anti- inflammatory factors. Most of the short and long-term complications of the neonatal sepsis are strictly related to inflammatory mediators. Neonatal sepsis is associated with a mortality rate that ranges from 13 to 60% inspite of improved antibiotic therapy and an increased morbidity in survivors .

DETAILED DESCRIPTION:
"Suspected sepsis" is one of the most frequently encountered diagnosis in neonatology because: a) a large number of newborns are evaluated for early or late sepsis based on risk factors and for fear of missing a correct diagnosis and a prompt treatment ; b) in neonates, the clinical signs of infection are not specific, late, and the differential diagnosis with neonatal respiratory distress syndrome, aspiration syndromes or neonatal maladaptation to extra-uterine life is difficult ; c) blood culture - the golden standard in neonatal sepsis diagnosis - provides late information, has a poor accuracy, and is not universally available; and d) up to date, there is no an ideal diagnostic tool for neonatal infection . Therefore, diagnosis of neonatal sepsis is still a challenge for neonatal medicine.

Antibiotic therapy is often initiated based upon clinical suspicion and/or the presence of risk factors, leading to excessive antibiotic therapy. Very often the diagnosis criteria for neonatal sepsis consists in documenting an infection in a newborn with severe systemic disease in which all possible noninfectious explanations for the patient's altered physiological status are either ruled out or unlikely.

The "gold standard", definitive test for neonatal sepsis is the isolation of the pathogen from blood. However, its accuracy is influenced by multiple factors a) contamination during sampling; b) sampling after antibiotic therapy was started; c) insufficient sampling volume; d) low colony count bacteremia. Accuracy of the blood culture varies between8 and 73% in various studies .

Despite hundreds of published studies, there is still no consensus regarding the best screening test or panel of tests for rapid detection of neonatal sepsis. Recently, new acute phase proteins, cytokines, cell surface antigens, and bacterial genome are used to improve the neonatal sepsis diagnosis but data are still under evaluation and most of these tests are either not clinically available or they are expensive .

Accumulating evidence indicates that the CBC is an effective predictor of prognosis and mortality in many disease states, including hematological disease, neoplasms, and severe infections. Therefore, non- specific changes in the CBC in critically ill neonates could be considered a key prognostic factor in the evaluation of survival prediction in these patients .

Some prognostic scoring systems with performance status, clinical symptoms and biochemical parameters help to guide accurate prediction of the prognosis, such as the acute physiology and chronic health evaluation, yet are considered too complex for general clinical use. Therefore, the prediction of clinical events with laboratory parameters, including complete blood cell count (CBC), has become an increased focus of research .

Total leukocyte count (TLC), total neutrophil count, ANC, immature neutrophil count, immature/total neutrophil ratio (I:T ratio), immature/mature neutrophil ratio (I:M ratio), neutrophil degenerative changes (vacuolization, toxic granulations, and Döhle bodies), and platelet count are the most used hematological parameters for Early Onset Sepsis evaluation . Most of the hematological screening panels for Early Onset Sepsis use a total leukocyte count < 5000 cells/mm3 or > 20.000 cells/mm3, an I:T ratio > 0.2, and total outside the normal range. TLC increases in severe neonatal infections (both mature and immature cells) possible secondary to growth factors and cytokine release that stimulate the bone marrow production.

Thrombocytopenia is one of the early but non-specific indicator of neonatal sepsis with or without DIC. It can be caused by bacterial, viral, fungal and parasitic infections and other non-infectious causes. The overall prevalence of thrombocytopenia in neonatal age group varies from1- 5%, and is reported to be much higher in newborns admitted to intensive care units, i.e. ranging from 22% to 35%. Severe thrombocytopenia (50000/mm3) was found to be present in 2.4% patients admitted in NICU.Bleeding is a major complication of thrombocytopenia but is generally limited to infants with count< 30000/mm3. Studies have shown that approximately 50% cases of culture proven of sepsis get thrombocytopenia .Changes in other platelet indices, like MPV(mean platelet volume) and PDW (platelet distribution width) have also been examined in relationship to neonatal sepsis in some studies .

Platelet indices (platelet counts, platelet distribution width-(PDW), mean platelet volume (MPV)) are one such set of parameters which can be helpful for the diagnosis and hence early treatment of neonatal sepsis. Advantages of platelet indices are that the sample for these can be drawn at the same time as that for other investigations and require no special sampling techniques and are easily available. Some studies had reported a low platelet counts, high mean platelet volume and platelet distribution width was observed in sepsis cases with a statistically significant difference as compared to controls .

ELIGIBILITY:
Inclusion Criteria:

1. Neonates with suspected sepsis that show non-specific signs and symptoms or focal signs of infection, including temperature instability, hypotension, poor perfusion with pallor and mottled skin, metabolic acidosis, tachycardia or bradycardia, apnoea, respiratory distress, grunting, cyanosis, irritability, lethargy, seizures, feeding intolerance, abdominal distention, jaundice, petechiae, purpura, and bleeding. Later complications of sepsis might include respiratory failure, pulmonary hypertension, cardiac failure, shock, renal failure, liver dysfunction, cerebral edema or thrombosis, adrenal hemorrhage or insufficiency, bone marrow dysfunction (neutropenia, thrombocytopenia, anemia), and disseminated intravascular coagulation.
2. Cases with neonatal sepsis diagnosed by isolating the causative agent from a normally sterile body site (blood, CSF, urine, pleural, joint, and peritoneal fluids (Andi L Shaneetal, 2017).

Exclusion Criteria:

1. Obvious features of dehydration
2. Major congenital malformations.
3. GIT functional or organic obstruction, hematological disorders, hypersplenism, respiratory distress, malignancy and neurological emergency as intra cranial hemorrhage.
4. Hypoxic ischemic encephalopathy.
5. Post-surgical cases which need NICU observation.

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: newborns with neonatal sepsis
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-09-30 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
white blood cells | one year
  total leucocytic count
white blood cells indices | one year
  total neutrophil count
Platelets indices | one year
  Platelet count
Platelets indices | one year
  Platelet distribution width(PDW)
Platelets indices | one year
  Mean platelet volume

CONTACTS AND LOCATIONS:
Overall Officials: Eslam A Roshdy, Principal Investigator — Assiut University Faculty of Medicine
Locations (1):
- Eslam Ahmad Roshdy, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
all collected IPD